CLINICAL TRIAL: NCT01894854
Title: Evaluation of the Furlong Evolution Uncemented Hip Prosthesis With Special Emphasize on the Use of Collared Design or Not. A Prospective, Randomized Study Evaluated by RadioStereometric Analysis (RSA) and DXA.
Brief Title: RSA Study of Furlong Evolution With and Without Collar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: JRI Orthopaedics Ltd (Industry)
Responsible Party: Principal Investigator, Gunnar Flivik, Associate professor, MD PhD, Region Skane
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Furlong Evolution_EW
Record Dates: First submitted 2013-07-01; First posted 2013-07-10 (Estimated); Last update posted 2025-06-24 (Actual); Status verified 2025-04

CONDITIONS: Hip Replacement in Osteoarthritis Patients
Keywords: Radiostereometry; Total Hip Arthroplasty; Stem design

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stem collar (No Intervention): The stem has two versions, one with and one without a collar. This arm will have stems with a collar. The classical Furlong HAC had a collar.
- No Stem collar (Active Comparator): The stem has two versions, one with and one without a collar. This arm will have stems without a collar. The classical Furlong HAC had a collar.
  Interventions: Procedure: Stem collar

INTERVENTIONS:
Procedure: Stem collar — The stem has two versions, one with and one without a collar. The classical Furlong HAC had a collar.
  Other Names: Furlong Evolution with collar; Furlong Evolution without collar
  Arms: No Stem collar

SUMMARY:
The aim of this study is to further investigate the clinical and radiological importance of design changes in cementless hip prosthesis. The investigators have earlier evaluated the classical Furlong HAC total hip prosthesis and a first design change Furlong Active. Now a further development, Furlong Evolution, is to be evaluated. This prosthesis, furthermore, comes with and without a collar, and the investigators are going to randomize between the two. The investigators hypothesize that the new design will be easier to implant and will present equal or less migration than the older designs which would imply a favourable outcome in the long term. The investigators further hypothesize that the collar play no major part for the long term migration and bone remodelling.

We will now do a 10 year follow up of the patients including RSA, DXA and PROMS

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of the hip necessitating primary hip replacement
* A femur considered suitable for uncemented fixation of the stem
* Biological age <75 years old at the inclusion time of the study.

Exclusion Criteria:

* Rheumatoid arthritis
* Malignant disease
* Severe osteoporosis
* Earlier fracture or operation in the hip to be operated on
* Peroperative fracture
* Ongoing corticosteroid (oral) or immunosuppressive medication
* Personal disorders (dementia, alcohol or drug abuse etc) suspected of making completion of the trial uncertain.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2025-03 (Actual)

PRIMARY OUTCOMES:
Radiostereometric Analysis (RSA) | The first postoperative day, 14 days, 3 months, 1, 2, 5 and 10 years
  This will measure the change in migration (translation and rotation around the x-, y-, and z-axis of the hip) over time. The migration pattern the first 2 years can predict the long term outcome.

SECONDARY OUTCOMES:
Dual-energy X-ray absorptiometry (DXA) | 14 days postoperatively and after 1, 5 and 10 years
  This will measure the change in bone density around the prosthesis during the first important year. This will tell if there is a bone resorption around the stem or cup.
General health questionnaire | Preoperatively (3-4 weeks) and 1, 2, 5 and 10 years postoperatively
  EuroQol (EQ-5D) - a standardized instrument for use as measure of general health outcome over time
Hip specific health questionnaire | Preoperatively (3-4 weeks) and 1, 2, 5 and 10 years postoperatively
  Hip disability and Osteoarthritis Outcome Score (HOOS) - this is a hip specific questionnaire that will measure how the operation has affected the patients function and pain situation.

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Flivik, MD PhD, Principal Investigator — Dept of Orthopedics, Skane University Hospital, Lund University, Sweden
Locations (1):
- Department of Orthopedics, Skane University Hospital, Lund University, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belfrage O, Weber E, Sundberg M, Flivik G. Preserved periprosthetic bone stock at 5 years post-operatively with uncemented short hip stem in both collared and collarless version. Arch Orthop Trauma Surg. 2022 Nov;142(11):3489-3496. doi: 10.1007/s00402-021-04225-z. Epub 2021 Nov 29. PMID 34841462